CLINICAL TRIAL: NCT05867745
Title: Evaluation of the Development of the Burdett National Transition Nursing Network
Brief Title: The National Transition Evaluation Study
Acronym: NTES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Surrey (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Burdett Trust for Nursing (Other); Imperial College Healthcare NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Somerset NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SPON 2022 05 FHMS; 313576 (Other: IRAS number)
Record Dates: First submitted 2023-04-28; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Young People With All Long-term Health Conditions
Keywords: young people; parents; transition into adult services; long-term health conditions
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lead nurse for Transition/Regional Nurse Advisors: The Lead Nurse and RNAs will be interviewed using telephone or online via Zoom. The interviews will be recorded using a Dictaphone rather than being saved via Zoom. Recordings will then be saved on the University's secure, password protected SharePoint for the study. Only the research team, and the designated transcriber, will have access to interview data. At the start of the project, interviews have been conducted in a PPI format to explore in depth the programme, expectations of how it should work and its implementation in order for the research team to devise the study. For the purposes of the research, interviews will be undertaken at one year, two years, and at the end of the programme to further explore implementation of the programme, including what works well, challenges encountered and their perceptions of the impact the programme has on families' experiences.
  Interventions: Other: Interview
- Young people: Young people aged 12 to 25 years will be invited to participate. Young people will be asked to complete surveys at baseline, six months to one year and 18 months.
  Survey: Online surveys (Qualtrics) will be used to collect data from young people participating in the case studies. Young people will be asked to provide basic demographic details: age, gender, health condition, and type of service they attend (children's/young person's/adults') and length of time since transfer to adult services (if already transitioned).
  Letter/email/video to a friend: Young people will also be asked to write a 'letter/email to a friend' to describe their experiences. This will be completed online with the survey. They will be invited to write a letter/email or record a video about a recent clinic appointment/encounter with a health professional.
  Interventions: Other: Survey; Other: Letter to a friend (autoethnography)
- Parents: Case study: Parents/carers will be invited to participate alongside young people. We will aim transition (including preparation, transfer and within adult services). Survey: Parents/carers of young people participating in the case study will be invited to complete an online survey (Qualtrics). Basic demographic details will be requested about the parent: age and gender; and their child: age, gender, health condition, and type of service they attend (children's/young person's/adults'), length of time since transfer to adult services (if already transitioned).
  Letter/email/video about their experiences: Parents will also be asked to complete a written task/video. They will be asked to describe their experiences relating to the shift in responsibility towards their child as the primary partner in their own healthcare, how their child is moving (or has moved) towards greater independence and competence in self-management.
  Interventions: Other: Survey; Other: Letter to a friend (autoethnography)
- Transition champions/key professionals: Transition champions and key professionals in participating Trusts who are involved in the care of young people included in the case studies will be identified by the RNAs. We will aim to involve staff from various professional roles. They will be invited to complete an online survey (using Qualtrics) during the first year and one at the end of the second year, towards the end of the project. The surveys will explore their views on the implementation of the programme, experiences of building/making changes to a transition service, including what works well, challenges encountered and their perceptions of the impact the programme has on families' experiences. One professional from each case study site will be interviewed via Zoom/telephone to explore these aspects more in-depth at the same time points as the surveys. Ideally, we will aim to interview the same professionals at both time points. Data access and storage for will be the same as for the Lead Nurse/RNA interviews.
  Interventions: Other: Interview; Other: Survey

INTERVENTIONS:
Other: Interview — As previously specified
  Groups: Lead nurse for Transition/Regional Nurse Advisors; Transition champions/key professionals
Other: Survey — As previously specified
  Groups: Parents; Transition champions/key professionals; Young people
Other: Letter to a friend (autoethnography) — As previously specified
  Groups: Parents; Young people

SUMMARY:
This is a multi-centre study within England to evaluate whether the Burdett Trust National Transition Network and the implementation of the Model of Improvement for Transition has an impact on the experience of transitioning from child to adult services for young people, and their families. A concurrent mixed methods design will be utilised with qualitative (interviews/case studies), and quantitative descriptive (surveys) data collected simultaneously over three phases. Participants will include young people, parents, and professionals involved in the young person's transition journey.

DETAILED DESCRIPTION:
This study forms the evaluation aspect to a large transition-related innovation that is taking place across England (https://www.leedsth.nhs.uk/burdett-national-transition-nursing-network/).

It is important to formally evaluate this process. The study has been designed to determine whether the Burdett National Transition Network and implementation of the Model of Improvement for Transition has an impact on the experience of transitioning from child to adult services for young people, and their families. The research team at the University of Surrey will conduct a three-phased, mixed methods study to understand the experiences of all relevant stakeholders involved in the Network and the model's implementation and transition service users. The overall aim is to document new learning to ensure maximum reach of the model within a network of transition care, and improve the outcomes for young people transitioning to adult services.

STUDY DESIGN Our intention is to undertake a process evaluation using a case study approach. The investigators want to look at the change from before, during and after the Model of Improvement for Transition's implementation. The investigators plan to gather data at the start of the project about what happens now, and then what happens as the Model of Improvement for Transition evolves. The investigators will also gather information that is already routinely collected on an ongoing basis in each of the sites working with the RNAs, as part of the overall implementation project. This will be provided in summary form. As this is an evolving process, this may include but may not be limited to the:

1. Number of Transition Lead roles for a whole organisation;
2. Number of organisations working through Transition QI process;
3. Number of organisations with transition contact;
4. Number of organisations with an Executive Lead for transition;
5. Number of Quality Improvement (QI) transition pathways completed;
6. Number of health-based youth workers that are in post to support transition;
7. Number of organisations with processes in place to use feedback from young people to support service improvement;
8. Number of organisations with effective Transition governance processes in place e.g. transition board, steering group, organisational policy and reporting.

Two organisations or services per region (eight study sites in total) that is involved in the transition of young people to adult health services will be selected as case studies, giving eight case studies in total. To inform an unbiased selection of cases, a list of criteria will be described a priori by the project team, a consensus will be reached on the type, and context of the services to be included based on maximum variation, for example, geography and deprivation score, size of institution or service, ethnic diversity of the population, type of long-term health condition. The investigators aim to include populations that are under-researched such as: young people with complex needs, mental health problems, looked after children, young people receiving palliative care, and those for whom English is not their first language.

THEORETICAL FRAMEWORK

The 'On Your Own Feet Ahead' framework provides a focus for our study. The framework addresses eight key elements of good transitional care, divided into three core categories:

1. interventions to improve the organisation of care;
2. interventions to stimulate independence and self-management of young people, and
3. collaboration with young people (and their families) and within the multidisciplinary team of professionals, working both in child and adult health care.

METHODS

It is well recognised that the most challenging aspect of changing practice is implementation and 'normalisation' of the 'intervention': therefore both qualitative (interviews) and quantitative descriptive (surveys) will have an important role to play in gathering contextual information from staff regarding how the Model of Improvement for Transition is both received and delivered. In order to understand the context and how the Model of Improvement for Transition is received and delivered our evaluation over three phases with repeated measures will include:

* The National Lead Nurse (Interviews)
* Regional Nurse Advisors (Interviews)
* Transition champions the Regional Nurse Advisors work with in the Trusts and key professionals in the various networks (case studies; survey/interviews)
* Young people and their parents/carers (case studies: survey/letter to a friend)

DATA ANALYSIS Survey data will be exported from Qualtrics to SPSS for analysis. Data stored within Qualtrics will be deleted upon study completion. Participants will be given a unique study ID. Only the study team will know the identity of the participants, necessary for the integration and synthesis of the survey and letter to a friend data or interview data. Survey data quality will be assessed for item/scale missingness at each time point and handled in accordance with scale guidelines (where available). Survey data will be analysed using descriptive statistics (e.g., means (standard deviations), medians (interquartile range) for continuous data, frequencies for categorical data) and presented by key group characteristics where appropriate (e.g., age group, gender etc) If appropriate, changes in the measurements over time will be tested with two-tailed, paired sample T-tests and Wilcoxon Matched Pair Signed Rank tests (Transition champion/key professionals), and repeated measures ANOVA (young people and parents) . Statistical significance will be considered at p ≤0.05 and as an exploratory study no adjustments will be made for multiple comparisons.

Interviews with the RNAs and Lead Nurse will be transcribed for analysis by a transcription company approved by the University of Surrey. The confidentiality agreement is provided with this application and can be found in clause 15 of the Transcription purchase order terms and conditions document. Any identifying information (e.g. names of people/hospitals) will be removed from the transcripts by the Researcher following transcription. The interviews will be analysed using thematic analysis.

The narratives in videos from the letter/email/video to a friend activity will be analysed using qualitative content analysis. The videos will not be transcribed. The research team will develop a proforma for the parents' videos and a separate one for young people's videos. Proformas will be developed by the researchers watching two videos each and coming together to discuss the elements of the video. These proformas will be used for analysis of subsequent videos.

Study data will be stored within SharePoint on the University of Surrey's password protected server. Any files containing participant details will be password protected. Data will only be accessible to the research team at the University of Surrey.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged 12 to 25 years (upper age limit determined during the mapping and their parents/carers)
* Young people with any long-term health condition(s) that will require transfer to adult health care services and their parents/carers
* Young people who have already transferred to adult health care services within the last two years (at the point of recruitment) and their parents/carers
* The Lead Nurse for Transition and Regional Nurse Advisors directly involved in implementation of National Transition Network and the Model of Improvement for Transition
* Transition champions and key professionals involved in the young person's transition from child to adult services from the eight services/organisations which from the case study sites

Exclusion Criteria:

• Young people and parents/carers who the clinical team caring for them consider it not appropriate to invite them to participate.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Young people and parents/carers from the eight case study sites for this project are eligible to participate. Dyads of young people and parents will be invited to participate. In cases where either the parent or young person does not wish to take part, the other can still participate.
  The Lead Nurse for Transition and RNAs are eligible to participate due to their direct role in implementing the National Transition Network and the Model of Improvement for Transition.
  Transition champions and key professionals from the eight case study sites for this project are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate processes and outcomes, and to evaluate the reach of the Model of Improvement for Transition for young people transitioning from child into adult services, increases over time will be demonstrated in: | 2.5 years
  The number of Transition Lead roles for a whole organisation
The investigators expect to see an increase in: | 2.5 years
  The number of organisations working through Transition QI process
The investigators expect to see an increase in: | 2.5 years
  The number of organisations with transition contact
The investigators expect to see an increase in: | 2.5 years
  The number of organisations with an Executive Lead for transition
The investigators expect to see an increase in: | 2.5 years
  The number of Quality Improvement (QI) transition pathways completed
The investigators also expect to see an increase in: | 2.5 years
  The number of health-based youth workers that are in post to support transition
Lastly, The investigators also expect to see an increase in: | 2.5 years
  The number of organisations with processes in place to use feedback from young people to support service improvement

CONTACTS AND LOCATIONS:
Overall Officials: Faith Gibson, PhD, Principal Investigator — The University of Surrey/Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Derian House Children's Hospice, Chorley, Lancashire
  - Darent Valley Hospitals; Dartford and Gravesham NHS Foundation Trust, Dartford
  - Imperial College Healthcare NHS Trust, London
  - Oxleas NHS Foundation Trust, London
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at present

REFERENCES:
- [Derived] Porter L, Gibson F, Aldiss S, Morgan S, Stanton A, Carney S, Farooq A, Barlow I, Sultan H, Sipanoun P. Bringing Young People, Health and Social Care Professionals, Transition Champions and Policymakers Together Through Hybrid Methods of Participation: Creating a Space for Shared Understanding of What Is Required to Improve Young People's Healthcare Transition. Health Expect. 2025 Feb;28(1):e70136. doi: 10.1111/hex.70136. PMID 39888226
- [Derived] Sipanoun P, Aldiss S, Porter L, Morgan S, Powell E, Gibson F. Transition of young people from children's into adults' services: what works for whom and in what circumstances - protocol for a realist synthesis. BMJ Open. 2024 Jan 4;14(1):e076649. doi: 10.1136/bmjopen-2023-076649. PMID 38176872